CLINICAL TRIAL: NCT00100802
Title: A Phase II Study of Concurrent Radiation and Temozolomide Followed By Temozolomide and CCNU in the Treatment of Children With High-Grade Glioma
Brief Title: Radiation Therapy, Temozolomide, and Lomustine in Treating Young Patients With Newly Diagnosed Gliomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACNS0423; NCI-2012-02645 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ACNS0423; CDR0000407744; COG-ACNS0423; ACNS0423 (Other: Children's Oncology Group); ACNS0423 (Other: CTEP); U10CA098543 (NIH)
Record Dates: First submitted 2005-01-06; First posted 2005-01-07 (Estimated); Results first posted 2017-01-13 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Anaplastic Astrocytoma; Central Nervous System Neoplasm; Glioblastoma; Gliosarcoma; Spinal Cord Neoplasm
MeSH Terms: conditions — Astrocytoma; Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma; Spinal Cord Neoplasms | interventions — Lomustine; Radiotherapy; Radiation; Temozolomide

ARMS (1):
- Treatment (lomustine, temozolomide, radiation therapy) (Experimental): Patients receive oral temozolomide once daily on days 1-42. Patients also undergo concurrent radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33 and 36-40. Patients who did not undergo prior gross total resection also undergo boost radiotherapy once daily on days 43-47. Four weeks after completion of chemoradiotherapy, patients receive oral temozolomide once daily on days 1-5 and oral lomustine on day 1. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Lomustine; Radiation: Radiation Therapy; Drug: Temozolomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Lomustine — Given PO
  Other Names: 1-(2-Chloroethyl)-3-cyclohexyl-1-nitrosourea; 1-Nitrosourea, 1-(2-chloroethyl)-3-cyclohexyl-; Belustin; Belustine; CCNU; Cecenu; CeeNU; Chloroethylcyclohexylnitrosourea; Citostal; Gleostine; Lomeblastin; Lomustinum; Lucostin; Lucostine; N-(2-Chloroethyl)-N'-cyclohexyl-N-nitrosourea; Prava; RB-1509; WR-139017
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac; TMZ

SUMMARY:
This phase II trial is studying how well giving radiation therapy together with temozolomide and lomustine works in treating young patients with newly diagnosed gliomas. Radiation therapy uses high energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as temozolomide and lomustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with temozolomide and lomustine after surgery may kill any remaining tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare event-free survival of pediatric patients with newly diagnosed high-grade gliomas treated with adjuvant radiotherapy and temozolomide followed by temozolomide and lomustine with historical controls.

II. Determine the toxicity of this regimen in these patients. III. Correlate MGMT and p53 expression in tumor tissue with outcome in patients treated with this regimen.

IV. Correlate polymorphisms in GSTP1, GSTM1 and GSTT1 genes and GSTP1 protein expression in tumors with survival in patients treated with this regimen.

OUTLINE: This is a pilot, multicenter study.

CHEMORADIOTHERAPY: Patients receive oral temozolomide once daily on days 1-42. Patients also undergo concurrent radiotherapy once daily on days 1-5, 8-12, 15-19, 22-26, 29-33 and 36-40. Patients who did not undergo prior gross total resection also undergo boost radiotherapy once daily on days 43-47.

MAINTENANCE CHEMOTHERAPY: Four weeks after completion of chemoradiotherapy, patients receive oral temozolomide once daily on days 1-5 and oral lomustine on day 1. Treatment repeats every 42 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year, every 6 months for 3 years and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, newly diagnosed high-grade glioma of 1 of the following histologies:

  * Anaplastic astrocytoma
  * Glioblastoma multiforme
  * Gliosarcoma
* Primary spinal cord malignant gliomas allowed
* No primary brainstem tumors
* Has undergone surgical resection or biopsy of the tumor within the past 31 days

  * Pre-operative and post-operative brain MRI with and without gadolinium-contrast OR pre-operative and post-operative spine MRI for spinal cord primaries

    * Post-operative MRI not required for patients who undergo biopsy only
* No evidence of neuraxis dissemination

  * Spine MRI and cerebrospinal fluid cytology required only if clinically indicated
* Performance status - Karnofsky 50-100% (for patients > 16 years of age)
* Performance status - Lansky 50-100% (for patients ≤ 16 years of age)
* At least 8 weeks
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8 g/dL (transfusions allowed)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN
* Albumin ≥ 2 g/dL
* Creatinine ≤ 1.5 times ULN
* Creatinine clearance or radioisotope glomerular filtration rate ≥ lower limit of normal
* No evidence of dyspnea at rest
* No exercise intolerance
* Pulse oximetry ≥ 94% (if determination is clinically indicated)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* Able to swallow oral medication
* Seizures allowed provided they are well controlled with anticonvulsants
* No hypersensitivity to temozolomide
* No prior biologic agents
* No prior chemotherapy
* Prior corticosteroids allowed
* No concurrent corticosteroids as an antiemetic
* Concurrent corticosteroids allowed only for treatment of increased intracranial pressure
* No concurrent radiotherapy using cobalt-60
* See Disease Characteristics
* No other prior treatment
* No concurrent phenobarbital or cimetidine
* No concurrent co-trimoxazole for Pneumocystis carinii pneumonia prophylaxis during study chemoradiotherapy

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 118 (Actual)
Dates: Start 2005-03-21 (Actual); Primary Completion 2012-09-01 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Regina I Jakacki, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Pollack IF, Hamilton RL, Burger PC, Brat DJ, Rosenblum MK, Murdoch GH, Nikiforova MN, Holmes EJ, Zhou T, Cohen KJ, Jakacki RI; Children's Oncology Group. Akt activation is a common event in pediatric malignant gliomas and a potential adverse prognostic marker: a report from the Children's Oncology Group. J Neurooncol. 2010 Sep;99(2):155-63. doi: 10.1007/s11060-010-0297-3. Epub 2010 Jul 4. PMID 20607350
- [Background] Pollack IF, Hamilton RL, Sobol RW, Nikiforova MN, Nikiforov YE, Lyons-Weiler MA, LaFramboise WA, Burger PC, Brat DJ, Rosenblum MK, Gilles FH, Yates AJ, Zhou T, Cohen KJ, Finlay JL, Jakacki RI; Children's Oncology Group. Mismatch repair deficiency is an uncommon mechanism of alkylator resistance in pediatric malignant gliomas: a report from the Children's Oncology Group. Pediatr Blood Cancer. 2010 Dec 1;55(6):1066-71. doi: 10.1002/pbc.22634. PMID 20589656
- [Result] Pollack IF, Hamilton RL, Sobol RW, Nikiforova MN, Lyons-Weiler MA, LaFramboise WA, Burger PC, Brat DJ, Rosenblum MK, Holmes EJ, Zhou T, Jakacki RI; Children's Oncology Group. IDH1 mutations are common in malignant gliomas arising in adolescents: a report from the Children's Oncology Group. Childs Nerv Syst. 2011 Jan;27(1):87-94. doi: 10.1007/s00381-010-1264-1. Epub 2010 Aug 20. PMID 20725730

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgery, Chemoradiotherapy, Rest, Maintenance, Follow-up: Patients must begin therapy within 31 days of surgery. Chemoradiotherapy = Radiation Therapy Dose: 54.0 Gy with a Boost of 5.4 Gy Temozolomide 90mg/m2/day daily for 42 days. Maintenance consists of 6 treatment cycles of combo chemotherapy with lomustine and temozolomide. Maintenance will begin 4 weeks following radiation. Five days of temozolomide (day 1 - 5) and one dose of lomustine (day 1) followed by 36 days of rest = 1 treatment cycle.
  lomustine: Capsule
  temozolomide: Capsule
  adjuvant therapy
  radiation therapy
Period: Overall Study
Arm/Group | Surgery, Chemoradiotherapy, Rest, Maintenance, Follow-up
Started | 118
Completed | 38
Not Completed | 80
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Lack of Efficacy | 47
Not completed — Physician Decision | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 5
Not completed — Ineligible | 12

BASELINE CHARACTERISTICS:
Groups:
- Surgery, Chemoradiotherapy, Rest, Maintenance, FUP: Patients must begin therapy within 31 days of surgery. Chemoradiotherapy = Radiation Therapy Dose: 54.0 Gy with a Boost of 5.4 Gy Temozolomide 90mg/m2/day daily for 42 days. Maintenance consists of 6 treatment cycles of combo chemotherapy with lomustine and temozolomide. Maintenance will begin 4 weeks following radiation. Five days of temozolomide (day 1 - 5) and one dose of lomustine (day 1) followed by 36 days of rest = 1 treatment cycle.
  lomustine: Capsule
  temozolomide: Capsule
  adjuvant therapy
  radiation therapy
Arm/Group | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP
Number analyzed (Participants) | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 110
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 12 [3 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55
  Male | 63
Region of Enrollment [Number; unit: participants]
  Canada | 15
  New Zealand | 1
  United States | 98
  Australia | 4

OUTCOME MEASURES:

1. Primary Outcome: One Year Overall Survival
Description: Estimated one year survival using the Kaplan-Meier methodology.
Time Frame: One year
Population: Population is based on 106 eligible patients out of 118 patients enrolled.
Measure: Number (95% Confidence Interval); unit: Estimated probability
Arm/Group | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP
Number analyzed (Participants) | 106
Estimated probability | 0.7208 [0.6237 to 0.7968]

2. Primary Outcome: Occurrence of Death Attributable to Complications of Protocol Therapy
Description: Number of deaths due to complications of protocol therapy.
Time Frame: While receiving protocol therapy (up to 301 days excluding delays) or within 30 days of Termination of Protocol Therapy
Population: 106 eligible patients out of 118 patients enrolled is the population basis for this outcome measure.
Measure: Number; unit: patients
Arm/Group | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP
Number analyzed (Participants) | 106
patients | 1

ADVERSE EVENTS:
Description: Serious adverse events, only eligible patients are considered. Other adverse events, only eligible patients are considered
Arm/Group | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP
Serious Adverse Events (participants affected / at risk) | 3/106
Other Adverse Events (participants affected / at risk) | 83/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP (N=106)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgery, Chemoradiotherapy, Rest, Maintenance, FUP (N=106)
Anemia (Blood and lymphatic system disorders) | 26 (26)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 (5)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Cushingoid (Endocrine disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Extraocular muscle paresis (Eye disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Papilledema (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (10)
Oral pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 10 (10)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Allergic reaction (Immune system disorders) | 2 (2)
Anorectal infection (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Gum infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 5 (5)
Meningitis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3)
Blood bilirubin increased (Investigations) | 4 (4)
GGT increased (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 36 (36)
Neutrophil count decreased (Investigations) | 59 (59)
Platelet count decreased (Investigations) | 56 (56)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 48 (48)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Abducens nerve disorder (Nervous system disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 7 (7)
Dysphasia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 5 (5)
Hydrocephalus (Nervous system disorders) | 3 (3)
IVth nerve disorder (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 3 (3)
Nervous system disorders - Other, specify (Nervous system disorders) | 3 (3)
Oculomotor nerve disorder (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Seizure (Nervous system disorders) | 8 (8)
Syncope (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Personality change (Psychiatric disorders) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (3)
Thromboembolic event (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.